CLINICAL TRIAL: NCT02056392
Title: A Phase I, Double-blind (Selumetinib [AZD6244; ARRY-142886] [Hyd-Sulfate]), Placebo-controlled, Open-Label (Moxifloxacin) Positive-controlled, Randomized, Three-period Crossover Study to Assess the Effects of Single Oral Dose of Selumetinib (75 mg) on QTc Interval Compared to Placebo, Using AVELOX (Moxifloxacin) as a Positive Control, in Healthy Male Volunteers Aged 18 to 45 Years
Brief Title: To Assess the Effects of Single Oral Dose of Selumetinib [AZD6244; ARRY-142886] [Hyd-Sulfate]), on QTc Interval in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D1532C00071
Record Dates: First submitted 2014-02-05; First posted 2014-02-06 (Estimated); Results first posted 2015-11-09 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-09

CONDITIONS: Solid Tumours
Keywords: Phase I, healthy, pharmacokinetics
MeSH Terms: interventions — AZD 6244; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Selumetinib 75mg (Experimental): Volunteers will receive selumetinib 75mg administered by mouth, as a capsule
  Interventions: Drug: Selumetinib
- Moxifloxacin 400 mg (Active Comparator): Volunteers will receive moxifloxacin 400mg administered by mouth, as a capsule
  Interventions: Drug: Moxifloxacin
- Selumetinib 75mg placebo (Placebo Comparator): Volunteers will receive selumetinib 75mg placebo, administered by mouth, as a capsule.
  Interventions: Drug: selumetinib placebo

INTERVENTIONS:
Drug: Selumetinib — Volunteers will receive 75 mg selumetinib oral dose (Treatment A)
  Other Names: AZD6244
  Arms: Selumetinib 75mg
Drug: Moxifloxacin — Volunteers will receive 400 mg Moxifloxacin oral dose (Treatment B)
  Other Names: Avelox®
  Arms: Moxifloxacin 400 mg
Drug: selumetinib placebo — Volunteers will receive selumetinib placebo oral dose (Treatment C)
  Other Names: AZD6244 placebo
  Arms: Selumetinib 75mg placebo

SUMMARY:
Study to assess the effect of Selumetinib [AZD6244; ARRY-142886] [Hyd-Sulfate]), on QTc interval in healthy male volunteers.

DETAILED DESCRIPTION:
A double-blind (Selumetinib [AZD6244; ARRY-142886] [Hyd-Sulfate]), Placebo-controlled, Open-Label (Moxifloxacin) Positive-controlled, Randomized, Three-period Crossover Study to Assess the Effects of Single Oral Dose of Selumetinib (75 mg) on QTc Interval Compared to Placebo, using AVELOX (Moxifloxacin) as a Positive Control, in Healthy Male Volunteers

ELIGIBILITY:
Inclusion Criteria: 1. Have a body mass index (BMI) between 18 and 30 kg/m2 and weigh at least 50 kg and no more than 100 kg (inclusive). 2. Must have not smoked in the last 30 days prior to screening for this study. 3. Have a calculated creatinine clearance (CrCL) greater than 50 mL/min using the Cockcroft-Gault formula.

Exclusion Criteria: 1. Subjects of Japanese or non-Japanese Asian ethnicity. 2. Subjects where any one parent or grandparent (maternal or paternal) is Japanese or non-Japanese Asian (e.g. China, Taiwan, Korea, Philippines, Thailand, Vietnam, and Malaysia). Asian Indians are acceptable. 3. Past history of central serous retinopathy or retinal vein thrombosis,intraocular pressure greater than 21 mmHg or uncontrolled glaucoma. 4. Any clinically relevant abnormal findings in physical examination, hematology, clinical chemistry, urinalysis, vital signs or ECG at baseline in the opinion of the investigator. 5. History or presence of any clinically significant disease or disorder in the opinion of the investigator.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2014-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Rasmussen, MD, Principal Investigator — Quintiles 6700 W 115th Street, Kansas, US
Locations (1):
- Research Site, Overland Park, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Selumetinib/Moxifloxacin/Selumetinib Placebo | Moxifloxacin/Selumetinib/Selumetinib Placebo | Moxifloxacin/Selumetinib Placebo/Selumetinib | Selumetinib Placebo/Moxifloxacin/Selumetinib | Selumetinib Placebo/Selumetinib/Moxifloxacin | Selumetinib/Selumetinib Placebo/Moxifloxacin
Started | 10 | 9 | 9 | 9 | 8 | 9
Completed | 8 | 8 | 6 | 9 | 7 | 9
Not Completed | 2 | 1 | 3 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 2 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Selumetinib/Moxifloxacin/Selumetinib Placebo | Moxifloxacin/Selumetinib/Selumetinib Placebo | Moxifloxacin/Selumetinib Placebo/Selumetinib | Selumetinib Placebo/Moxifloxacin/Selumetinib | Selumetinib Placebo/Selumetinib/Moxifloxacin | Selumetinib/Selumetinib Placebo/Moxifloxacin | Total
Number analyzed (Participants) | 10 | 9 | 9 | 9 | 8 | 9 | 54
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26 (7) | 25 (5) | 25 (4) | 31 (8) | 28 (8) | 30 (9) | 27 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 10 | 9 | 9 | 9 | 8 | 9 | 54
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 7 | 5 | 4 | 4 | 5 | 4 | 29
  Black or African American | 3 | 4 | 5 | 5 | 3 | 5 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in QTcF
Description: Change from baseline in QTcF at 30 minutes (msec)
Time Frame: 30 min
Population: All patients who had evaluable pharmacodynamic data available for at least one treatment group were included in the PD analysis set
Measure: Least Squares Mean (95% Confidence Interval); unit: msec
Units Other Than Participants: change from baseline
Groups:
- Moxifloxacin: Moxiflxacin 400 mg (open label)
- Placebo: Selumetinib placebo (3 capsules)
- Selumetinib: Selumetinib 75mg bs (3x25mg capsules)
Arm/Group | Moxifloxacin | Placebo | Selumetinib
Number analyzed (Participants) | 50 | 49 | 50
Number analyzed (change from baseline) | 50 | 49 | 50
msec | 2.0 [0.5 to 3.5] | -4.1 [-5.6 to -2.5] | -4.2 [-5.7 to -2.7]
Statistical Analysis 1: Comparison: Placebo vs Selumetinib; 47 evaluable volunteers gives 90% power to show non-inferiority of selumetinib versus placebo across all 10 post-dose time points, using paired T-test, 1-sided alpha=0.05 and assuming a true difference of 3 msec; Test type: Non-Inferiority or Equivalence — All one-sided 95% confidence intervals at each time point for the selumetinib difference versus placebo (2-sided 90% CIs) should be less than 10ms; Mixed Models Analysis; Mean Difference (Final Values) = -0.2, 90% CI 2-sided [-1.8 to 1.5]
Statistical Analysis 2: Comparison: Moxifloxacin vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Mean Difference (Final Values) = 6.1, 90% CI 2-sided [4.4 to 7.7]

2. Primary Outcome: Change From Baseline in QTcF
Description: Change from baseline in QTcF at 1 hour (msec)
Time Frame: 1 hour
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: msec
Units Other Than Participants: change from baseline
Arm/Group | Moxifloxacin | Placebo | Selumetinib
Number analyzed (Participants) | 50 | 49 | 50
Number analyzed (change from baseline) | 50 | 49 | 50
msec | 7.9 [6.4 to 9.4] | -1.4 [-2.9 to 0.2] | -1.7 [-3.2 to -0.2]
Statistical Analysis 1: Comparison: Placebo vs Selumetinib; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Mean Difference (Final Values) = -0.4, 90% CI 2-sided [-2.0 to 1.3]
Statistical Analysis 2: Comparison: Moxifloxacin vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Mean Difference (Final Values) = 9.2, 90% CI 2-sided [7.6 to 10.8]

3. Primary Outcome: Change From Baseline in QTcF
Description: Change from baseline in QTcF at 1 hour 30 min (msec)
Time Frame: 1 hour 30 min
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: msec
Units Other Than Participants: change from baseline
Arm/Group | Moxifloxacin | Placebo | Selumetinib
Number analyzed (Participants) | 50 | 49 | 50
Number analyzed (change from baseline) | 50 | 49 | 50
msec | 8.1 [6.6 to 9.6] | -1.8 [-3.3 to -0.2] | -0.9 [-2.4 to 0.6]
Statistical Analysis 1: Comparison: Placebo vs Selumetinib; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Mean Difference (Final Values) = 0.9, 90% CI 2-sided [-0.7 to 2.5]
Statistical Analysis 2: Comparison: Moxifloxacin vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Mean Difference (Final Values) = 9.9, 90% CI 2-sided [8.3 to 11.5]

4. Primary Outcome: Change From Baseline in QTcF
Description: Change from baseline in QTcF at 2 hours (msec)
Time Frame: 2 hours
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: msec
Units Other Than Participants: change from baseline
Arm/Group | Moxifloxacin | Placebo | Selumetinib
Number analyzed (Participants) | 50 | 49 | 50
Number analyzed (change from baseline) | 50 | 49 | 50
msec | 7.9 [6.4 to 9.4] | -2.3 [-3.8 to -0.7] | -1.9 [-3.4 to -0.4]
Statistical Analysis 1: Comparison: Placebo vs Selumetinib; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Mean Difference (Final Values) = 0.4, 90% CI 2-sided [-1.2 to 2.0]
Statistical Analysis 2: Comparison: Moxifloxacin; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Mean Difference (Final Values) = 10.1, 90% CI 2-sided [8.5 to 11.8]

5. Primary Outcome: Change From Baseline in QTcF
Description: Change from baseline in QTcF at 3 hours (msec)
Time Frame: 3 hours
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: msec
Units Other Than Participants: change from baseline
Arm/Group | Moxifloxacin | Placebo | Selumetinib
Number analyzed (Participants) | 50 | 49 | 50
Number analyzed (change from baseline) | 50 | 49 | 50
msec | 8.8 [7.3 to 10.3] | -3.2 [-4.7 to -1.6] | -3.3 [-4.8 to -1.8]
Statistical Analysis 1: Comparison: Placebo vs Selumetinib; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Mean Difference (Final Values) = -0.2, 90% CI 2-sided [-1.8 to 1.5]
Statistical Analysis 2: Comparison: Moxifloxacin vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Mean Difference (Final Values) = 11.9, 90% CI [10.3 to 13.6]

6. Primary Outcome: Change From Baseline in QTcF
Description: Change from baseline in QTcF at 4 hours (msec)
Time Frame: 4 hours
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: msec
Units Other Than Participants: change from baseline
Arm/Group | Moxifloxacin | Placebo | Selumetinib
Number analyzed (Participants) | 50 | 49 | 50
Number analyzed (change from baseline) | 50 | 49 | 50
msec | 8.6 [7.1 to 10.1] | -2.2 [-3.7 to -0.7] | -3.7 [-5.2 to -2.2]
Statistical Analysis 1: Comparison: Placebo vs Selumetinib; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Mean Difference (Final Values) = -1.5, 90% CI 2-sided [-3.1 to 0.2]
Statistical Analysis 2: Comparison: Moxifloxacin vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Mean Difference (Final Values) = 10.8, 90% CI 2-sided [9.2 to 12.5]

7. Primary Outcome: Change From Baseline in QTcF
Description: Change from baseline in QTcF at 6 hours (msec)
Time Frame: 6 hours
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: msec
Units Other Than Participants: change from baseline
Arm/Group | Moxifloxacin | Placebo | Selumetinib
Number analyzed (Participants) | 50 | 49 | 50
Number analyzed (change from baseline) | 50 | 49 | 50
msec | 4.7 [3.2 to 6.2] | -4.1 [-5.6 to -2.6] | -5.9 [-7.4 to -4.4]
Statistical Analysis 1: Comparison: Placebo vs Selumetinib; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Mean Difference (Final Values) = -1.8, 90% CI 2-sided [-3.4 to -0.1]
Statistical Analysis 2: Comparison: Moxifloxacin vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Mean Difference (Final Values) = 8.8, 90% CI 2-sided [7.1 to 10.4]

8. Primary Outcome: Change From Baseline in QTcF
Description: Change from baseline in QTcF at 8 hours (msec)
Time Frame: 8 hours
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: msec
Units Other Than Participants: change from baseline
Arm/Group | Moxifloxacin | Placebo | Selumetinib
Number analyzed (Participants) | 50 | 49 | 50
Number analyzed (change from baseline) | 50 | 49 | 50
msec | 3.6 [2.1 to 5.1] | -5.3 [-6.8 to -3.7] | -6.5 [-8.0 to -5.0]
Statistical Analysis 1: Comparison: Placebo vs Selumetinib; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Mean Difference (Final Values) = -1.3, 90% CI 2-sided [-2.9 to 0.4]
Statistical Analysis 2: Comparison: Moxifloxacin vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Mean Difference (Final Values) = 8.9, 90% CI 2-sided [7.2 to 10.5]

9. Primary Outcome: Change From Baseline in QTcF
Description: Change from baseline in QTcF at 12 hours (msec)
Time Frame: 12 hours
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: msec
Units Other Than Participants: change from baseline
Arm/Group | Moxifloxacin | Placebo | Selumetinib
Number analyzed (Participants) | 50 | 49 | 50
Number analyzed (change from baseline) | 50 | 49 | 50
msec | 4.2 [2.7 to 5.7] | -3.4 [-5.0 to -1.9] | -8.2 [-9.7 to -6.7]
Statistical Analysis 1: Comparison: Placebo vs Selumetinib; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Mean Difference (Final Values) = -4.7, 90% CI 2-sided [-6.4 to -3.1]
Statistical Analysis 2: Comparison: Moxifloxacin vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Mean Difference (Final Values) = 7.6, 90% CI 2-sided [6.0 to 9.3]

10. Primary Outcome: Change From Baseline in QTcF
Description: Change from baseline in QTcF at 24 hours (msec)
Time Frame: 24 hours
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: msec
Units Other Than Participants: change from baseline
Arm/Group | Moxifloxacin | Placebo | Selumetinib
Number analyzed (Participants) | 50 | 49 | 50
Number analyzed (change from baseline) | 50 | 49 | 50
msec | 2.4 [0.9 to 3.9] | -1.6 [-3.1 to -0.1] | -4.1 [-5.6 to -2.6]
Statistical Analysis 1: Comparison: Placebo vs Selumetinib; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Mean Difference (Final Values) = -2.5, 90% CI 2-sided [-4.1 to -0.9]
Statistical Analysis 2: Comparison: Moxifloxacin vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Mean Difference (Final Values) = 4.0, 90% CI 2-sided [2.4 to 5.7]

ADVERSE EVENTS:
Time Frame: AEs were collected for up to 5 weeks, this was from the day before the first randomised treatment period (Day -1, Visit 2) until the follow-up visit.
Description: Of the 54 participants in the study, 3 did not receive Selumetinib, 3 did not receive Moxifloxacin and 4 did not receive Selumetinib Placebo (due to discontinuing the study).
Arm/Group | Selumetinib | Moxifloxacin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/51 | 1/50
Other Adverse Events (participants affected / at risk) | 5/51 | 5/51 | 4/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Selumetinib (N=51) | Moxifloxacin (N=51) | Placebo (N=50)
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Selumetinib (N=51) | Moxifloxacin (N=51) | Placebo (N=50)
Headache (Nervous system disorders) | 3 | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less